CLINICAL TRIAL: NCT04550130
Title: An Open-label, Randomised, Multi-centre, Dose-Evaluation Study of the Efficacy and Safety of TLA Gut™ Leukapheresis Treatment in Patients With Ulcerative Colitis
Brief Title: Dose-Evaluation Study of the Efficacy and Safety of TLA Gut™ Leukapheresis Treatment in Patients With Ulcerative Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TLA, Targeted Immunotherapies AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLA002
Record Dates: First submitted 2020-04-09; First posted 2020-09-16 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low dose (1.8 L) (Experimental): Patients in this arm will be treated with one column (Leukapheresis) and 1.8 L blood will be filtered.
  Interventions: Device: TLA Gut™
- high dose (3.6 L) (Experimental): Patients in this arm will be treated with Two column (Leukapheresis) and 3.6 L blood will be filtered.
  Interventions: Device: TLA Gut™

INTERVENTIONS:
Device: TLA Gut™ — The medical device to be investigated is named Tailored Leukapheresis (TLA) Gut™. The device comprises a column that has been designed for extracorporeal leukapheresis to specifically remove chemokine (C-C motif) receptor 9 (CCR9) expressing immunological cell populations including human leukocyte antigen DR isotype (HLA-DRhi ) monocytes from the circulation. This is achieved by integrating a strong affinity binding between the gut homing cell receptor, CCR9, and its cognate ligand, thymus-expressed chemokine (TECK) or chemokine ligand 25 (CCL25). Those blood cells that express CCR9 will bind to presented Biotinylated thymus-engineered chemokine (bTECK) on the matrix by a strong receptor ligand interaction, remaining bound to the matrix. Blood cells that do not express the receptor pass through the column unchanged and are returned to the patient.

SUMMARY:
An open-label, randomised, multi-centre, dose evaluation study of the efficacy and safety of TLA Gut™ leukapheresis treatment in patients with UC. The aim of this trial is to evaluate the efficacy and safety of two different TLA Gut™ dose regimens in patients with acute exacerbation of UC. Enrolled patients will participate in a 6-week treatment phase and a 20- week follow-up phase. The treatment phase consists of two periods; 2 weeks in which patients will undergo two treatment sessions per week, followed by 4 weeks of a single treatment session per week. The follow-up phase consists of 2 visits, one visit at week 7 and the last visit at week 26. Telephone visits will be conducted between these visits. In all a patient will undergo 8 treatment visits and 2 follow-up visits. Only patients not having experienced an earlier recurrence will participate in the follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

Female or male patients 18 to 80 years of age

* Active UC without Ileorectal anastomosis (IRA)
* Active UC is defined as:

  * Total Mayo score of ≥ 6 to 11 points
  * Flexible rectosigmoidoscopy findings of 2 or 3 (0 inactive disease, 1; mild disease, 2; moderate disease or 3; severe disease)
* Minimum extension of inflammation 10 cm from anus.
* Active disease with no medical treatment OR Active disease despite receiving concomitant therapy with one or more of the following agents:

  * ≤20 mg prednisolone daily. Stable dose ≥1 week prior to the start of the investigation.
  * 5-Aminosalicylate (5-ASA) agents for ≥4 weeks and stable dose for ≥2 weeks (local or systemic administration)
  * Rectal administration of corticosteroids in a stable dose for ≥2 weeks
  * Azathioprine or 6-mercaptopurine for ≥8 weeks or stable dose ≥2 weeks
* No anti-tumour necrosis factor (TNF) treatment (Adalimumab, Infliximab, Golimumab, Certolizumab), anti-integrin-treatment (vedolizumab), Interleukin (IL)-12/23 inhibitor (Ustekinumab) or Janus Kinase (JAK) treatment (Tofacitinib) during the last 4 weeks prior to entering the study
* Patients with peripheral veins suitable for extracorporeal treatment - must be examined by the treating apheresis specialist
* Willing and able to give written informed consent

Exclusion Criteria:

Involvement in any investigational drug or device trial within 30 days prior to this investigation

* Patients with peripheral veins not suitable for extracorporeal treatment
* Fever, defined as a temperature of >38,5 Celsius degrees (ºC), at the Screening Visit
* Heart failure
* Coronary artery disease
* Cardiomyopathy
* Valvular heart disease
* Cardiac arrythmia class IV
* Underweight person (BMI < 19)
* Hypotension (< 90/55 mmHG)
* Hypoproteinemia
* Evidence of toxic megacolon
* History of hypersensitivity to heparin
* Heparin-induced thrombocytopenia
* History of cerebrovascular incident
* Known clinically significant bleeding disorder
* Colectomy planned within 6 months
* Concomitant anticoagulant therapy
* History of hypercoagulable disorders
* Severe anaemia or Leukopenia
* Patients with active viral hepatitis and/or human immunodeficiency virus (HIV) infections
* A positive urine pregnancy test at the screening visit
* Patients that are nursing Local intestinal treatments with suppositories, enemas, creams, ointments or foams during the last 2 weeks
* Current daily smoking habits
* Patients unwilling to meet the requirements of the clinical investigational plan
* Other medical or social reasons for exclusion at the discretion of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate whether the intervention of TLA Gut™ reduces Human Leukocyte Antigen DR isotype (HLADRhi) | baseline, during treatment (after 4 treatment sessions at week 2)
  Mean percentage change in HLA-DRhi expressing monocytes

SECONDARY OUTCOMES:
Evaluate the effect of intervention of TLA Gut™ on clinical, histopathology and laboratory criteria and variables | baseline, during treatment (after 4 treatment sessions at week 2)
  Mean change in HLA-DRhi expressing monocytes
Evaluate the effect of intervention of TLA Gut™ on clinical variables | baseline, after 4 treatment sessions at week 2 , immediately after treatment completion
  Mean change and mean percentage change in Mayo Score Index
Evaluate the effect of intervention of TLA Gut™ on laboratory criteria | baseline, during treatment (at week 6), immediately after treatment completion
  Mean percentage change in faecal calprotectin levels
Evaluate the effect of intervention of TLA Gut™ on clinical, histopathology and laboratory criteria and variables | immediately after treatment completion
  Proportion of patients in each dosing group achieving laboratory remission, clinical remission or both laboratory and clinical remission
Evaluate the effect of intervention of TLA Gut™ on clinical variables | immediately after treatment completion
  Proportion of patients in each dosing group classified as responders
Evaluate the effect of intervention of TLA Gut™ on clinical variables | baseline, after 4 treatment sessions at week 2 , immediately after treatment completion
  Mean change and mean percentage change in Mayo Endoscopic Sub-Score Index
Evaluate the effect of intervention of TLA Gut™ on clinical variables | baseline, after 4 treatment sessions at week 2 , immediately after treatment completion
  Mean change and mean percentage change in Ulcerative Colitis Endoscopic Index of Severity (UCEIS) score

CONTACTS AND LOCATIONS:
Locations (1):
- Ersta Sjukhus, Medicinkliniken, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No